CLINICAL TRIAL: NCT06917430
Title: Muscle MRI Outlining of Neuromuscular Diseases Using Artificial Intelligence
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bjørk Teitsdóttir, Stud.med, Rigshospitalet, Denmark
Other Study IDs: 115991
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Becker Muscular Dystrophy; FSHD - Facioscapulohumeral Muscular Dystrophy; Hypokalemic Periodic Paralysis
Keywords: AI; muscle delineation; automated segmentation; Becker muscular dystrophy; FSHD; HypoPP
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophy, Facioscapulohumeral; Hypokalemic Periodic Paralysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Becker muscular dystrophy: MRI scans
  Interventions: Other: No intervention
- HypoPP: MRI scans
  Interventions: Other: No intervention
- FSHD: MRI scans
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
Background and aim:

Neuromuscular diseases encompass a range of conditions affecting muscle cells, nerves, or the interaction between the two. A common pathological feature of these conditions is the pro-gressive replacement of muscle tissue with fat, which can be visualised using magnetic reso-nance imaging (MRI). MRI-based fat quantification serves as a key biomarker for disease characterisation, progression tracking, and treatment assessment. Currently, manual segmenta-tion of MRI scans for fat quantification is very time-consuming, requiring individual muscle delineation. Therefore, an artificial intelligence (AI) model is being developed to automate the segmentation. The aim of this study is to validate this AI model and assess its possibilities and limitations.

Method:

The study is ongoing. Retrospective MRI scans of patients with four different muscle diseases (anoctaminopathy, Becker muscular dystrophy, facioscapulohumeral muscular dystrophy, and hypokalemic periodic paralysis) are collected and manual delineation used for training the AI-model is being performed. The intramuscular fat fraction of individual muscles of the pelvis, thigh, and calf will be analysed using the AI model. The performance of the AI model will be compared to manual segmentation. The AI will be evaluated on metrics such as segmentation accuracy and time efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Genetically verified diagnosis of neuromuscular diseases.
* Age above 18 years

Exclusion Criteria:

* Contraindications to perform an MRI
* Competing disorders and other muscle disorders, which may alter measurements. The investigator will decide whether the competing disorder can significantly influence the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Copenhagen Neuromuscular Centre.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference in fat fraction between manual and AI outlining. | Analysis of the muscle fat fraction takes 1 hour per patient.
  The mean difference in MRI assessed intramuscular fat fraction in the lower back, thigh, and calf muscles between manual outlining and the outlining by the AI model.

SECONDARY OUTCOMES:
Correlation between Manual/AI outlining discrepancies and disease severity | The analysis of the MRI takes around an hour
  Investigate if the difference between manual outlining and AI outlining increases the more advanced stage the disease is. A correlation analysis will be made between manual/AI differences and fat fraction in lower back, thigh, and calf.

IPD SHARING:
Plan to Share IPD: Undecided